CLINICAL TRIAL: NCT04752085
Title: Prognosis and Course of COVID-19 Infection in Hospitalised Patients
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Olga Mironova, Associate Professor, I.M. Sechenov First Moscow State Medical University
Other Study IDs: 03-21
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: COVID-19; chitotriosidase; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Chitotriosidase activity — The chitotriosidase activity will be measured in all the subjects

SUMMARY:
The aim of the cohort prospective observational study is to define the major factors influencing the course of COVID-19 infections and its prognosis in hospitalised patients.

The investigators plan to include 300 patients hospitalised with COVID-19 infection.

The phone contacts with patients are due after 90 and 180 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalisation with COVID-19

Exclusion Criteria:

* History of hospitalisation with COVID-19 infection
* Discharge from the hospital before the end of the treatment course
* Transfer to another hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 patients hospitalised with COVID-19 infection
Sampling Method: Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Need in biological therapy or/and respiratory support | Up to 1 month
  The primary endpoint is the need in biological therapy or/and respiratory support including noninvasive ventilation during hospital stay

SECONDARY OUTCOMES:
Number of days spent in hospital | Up to 1 month
  The investigators plan to assess the overall length of hospitalisation due to COVID-19 infection as an outcome measure
All-cause death | 90 days
  To assess the all-cause death 90 days after discharge
All-cause death | 180 days
  To assess the all-cause death 180 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Olga Mironova, PhD, Principal Investigator — Sechenov University; Ekaterina Schelkanovtseva, MD, Study Chair — Sechenov University
Locations (2):
- Russia (2):
  - University Hospital #1, Moscow
  - University Hospital #4, Moscow

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schelkanovtseva ES, Isaev GO, Mironova OY, Balakhonov AA, Skvortsov AV, Nagornov IO, Suvorov AY, Fomin VV, Panferov AS. [The survival prediction of hospitalized patients with COVID-19: the role of chitotriosidase level in peripheral blood]. Ter Arkh. 2023 Sep 29;95(7):543-547. doi: 10.26442/00403660.2023.07.202280. Russian. PMID 38159003